CLINICAL TRIAL: NCT02076230
Title: A Phase I, Open-Label, Two-Center Trial to Investigate the Mass Balance and Metabolite Profile of TH-302 in Cancer Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 TH-302 Mass Balance Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200592-007; 2013-003950-25 (EudraCT Number)
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumor
Keywords: 14C-TH-302; Advanced or Metastatic Solid Tumors; Evofosfamide
MeSH Terms: interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- [14C] TH-302 (Label 1) (Experimental)
  Interventions: Drug: [14C] TH-302 (Label 1); Drug: Unlabeled TH-302
- [14C] TH-302 (Label 2) (Experimental)
  Interventions: Drug: [14C] TH-302 (Label 2); Drug: Unlabeled TH-302

INTERVENTIONS:
Drug: [14C] TH-302 (Label 1) — [14C]-labeled TH-302 (Label 1) will be administered as intravenous infusion over 30 minutes on Day 1 of Part A.
  Arms: [14C] TH-302 (Label 1)
Drug: [14C] TH-302 (Label 2) — [14C]-labeled TH-302 (Label 2) will be administered as intravenous infusion over 30 minutes on Day 1 of Part A.
  Arms: [14C] TH-302 (Label 2)
Drug: Unlabeled TH-302 — Unlabeled TH-302 will be administered along with labeled TH-302 at the dose of 340 milligram per square meter (mg/m^2) as intravenous infusion over 30 minutes on Day 1 of Part A, followed by recommended Phase 2 dose (RP2D) of 480 mg/m^2 as monotherapy infusion over 30 minutes on Days 8 and 15 of Part A; and on Days 1, 8 and 15 of Part B, until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow up, or death.

SUMMARY:
This is an open-label, Phase 1, two-center trial to evaluate the mass balance and metabolite profile of carbon 14 [14C]-labeled TH-302 (Label 1 and Label 2) followed by subsequent treatment with unlabeled TH-302 in cancer subjects with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male subject with pathologically or cytologically confirmed solid tumor which is locally advanced or metastatic, and either refractory to the standard therapy or for which no effective standard therapy is available
* Subject has measurable and evaluable disease as RECIST version 1.1
* Age greater than or equal to (>=) 18 years and less than or equal to (=<) 70 years
* Body mass index (BMI) >= 19 and =< 33 kilogram per square meter (kg/m^2), body weight greater than (>) 50 kilogram (kg)
* Eastern cooperative oncology group (ECOG) performance status of 0 to 1
* Life expectancy of at least 3 months
* At least 4 weeks from previous cytotoxic chemotherapy or radiation therapy and at least 5 half-lives or 6 weeks, whichever is longer, after targeted or biologic therapy
* Acceptable renal function, liver function and hematologic status as defined in the protocol
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* New York Heart Association (NYHA) Class 3 or 4 congestive heart disease, myocardial infarction within 6 months, unstable arrhythmia, symptomatic ischemic heart disease or symptomatic peripheral arterial vascular disease
* Severe chronic obstructive or other pulmonary disease with hypoxemia as defined in the protocol
* Major surgery, other than diagnostic surgery, =< 28 days prior to Day 1. Subject must have completely recovered from surgery
* Primary brain tumors or clinical evidence of active brain metastasis as defined in the protocol
* Treatment with strong inhibitors and/or inducers of drug metabolic enzymes or drug transporter as defined in the protocol
* Participation in a drug trial within 30 days prior to start of trial medication. Participation in a trial involving administration of 14C-labeled compound(s) within last 6 months prior to start of study drug
* Inability to understand the protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial
* Legal incapacity or limited legal capacity
* Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics profile in plasma: Cmax, Tmax, AUC (0-t), lambda_z, t1/2, AUC (0-infinity), CL, Vss, Vz, MRT for TH-302 and its active metabolite Br-IPM | Days 1 and 8 of Cycle 1
Pharmacokinetics profile in excreta: Cumulative Ae (0-t), Ae (0-infinity), percent radioactive dose excreted in urine and feces, AeUF, CLR, CLNR for TH-302 and its active metabolite Br-IPM | Day 1 of Cycle 1

SECONDARY OUTCOMES:
Number of subjects with Treatment-emergent adverse events (TEAEs) | Baseline up to Day 30 after the last dose of study treatment
Blood to plasma ratio of total 14C-radioactivity | Days 1 and 8 of Cycle 1
Total and free plasma concentrations of TH-302 in plasma | Day 1 of Cycle 1
Number of subjects with tumor response according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1) | Up to 1 year
  Tumor response was defined as the occurrence of complete response (CR) or partial response (PR) based on the investigator's assessment according to RECIST v 1.1.
Unbound fraction (fu) of TH-302 in plasma | Day 1 of Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center located in, Darmstadt, Germany